CLINICAL TRIAL: NCT05589402
Title: Temporary Inactivation of Strong Muscle Sensation to Improve Rehabilitation Interventions in SCI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Rio Grande Valley (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-18-0596
Record Dates: First submitted 2022-06-23; First posted 2022-10-21 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries; Spine Disease; Stroke
Keywords: Rehabilitation; Numbing; temporary deafferentation-induced cortical plasticity
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Diseases; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine Cream 5% (Experimental): A topical anesthetic will be used to deliver temporary inactivation of muscle sensation. Specifically, due to its high safety profile, Lidocaine Cream 5% will be used in the current sub-study. Lidocaine cream (5%) is FDA-approved and available over-the-counter. The investigators will apply the lidocaine cream 5% following FDA guidelines and previously published protocol methodology. A test will be utilized to evaluate if the approach provides complete and temporary inactivation of sensation from the biceps. The von Frey filament test will be used with filaments ranging in size (1,65 to 6,65) to be placed on the biceps muscle every 15 minutes after lidocaine application.
  Based on published work, and the current investigators' pilot data, it is anticipated that all sensations from the biceps should be blocked approximately 30 to 60 minutes after lidocaine application. Complete temporary inactivation will be defined at the point when all baseline sensation can no longer be achieved.
  Interventions: Drug: Lidocaine Cream 5%
- Rehabilitation Movement Training (Other): During temporary deafferentation, subjects will perform movement training. Similar to other single-session studies, the current investigators chose to pair the paradigm with movement training to bolster the effects of the approach.
  A reaching task that is commonly performed in rehabilitation will be used. Task practice will be performed for 1 hour, with breaks given every 10 minutes. Past experiments in the current investigators' lab have adopted a similar protocol for task practice in SCI and found no adverse events. Movement training will also be assisted by the Bionik InMotion Arm/Hand robot, which has been studied in clinical and rehabilitative practices for over 20 years.
  Movement training at 1 hour will be ceased due to issues with fatigue, as has been noted in previous SCI clinical studies. In addition, published work suggests that lidocaine has a half-life of one 1 hour. Thus, maximum benefits should be achieved at the 1-hour mark after application.
  Interventions: Other: Rehabilitation Movement Training

INTERVENTIONS:
Drug: Lidocaine Cream 5% — Ebanel 5% Lidocaine Topical Numbing Cream Maximum Strength 1.35 Oz, Numb520 Pain Relief Cream Anesthetic Cream Infused with Aloe Vera, Vitamin E, Lecithin, Allantoin, Secured with Child Resistant Cap
  Other Names: Ebanel; UBER NUMB
  Arms: Lidocaine Cream 5%
Other: Rehabilitation Movement Training — reaching tasks, hand exercises (e.g., putty, grip exerciser, resistance bands, etc).
  Arms: Rehabilitation Movement Training

SUMMARY:
The investigators are conducting a research study to try to improve rehabilitation interventions for individuals with spinal cord injury (SCI). In this study, the aim is to determine if temporarily numbing non-paralyzed arm muscles with an over-the-counter numbing cream while exercising paralyzed muscles, can improve the strength, function, and sensation of paralyzed muscles after a spinal cord injury.

DETAILED DESCRIPTION:
The functional benefits of temporary deafferentation (numbing)-induced cortical plasticity have been demonstrated in individuals with stroke, nerve damage, and pain syndromes. Of note, documented benefits have included improvements in motor function and touch perception in the weaker muscles. For example, Weiss et al demonstrated that temporary deafferentation to the forearm of the paretic limb in stroke for two hours during movement therapy improved motor performance of the hand by 10 to 48% after a single session. Another study established that bi-weekly sessions of temporary deafferentation for two weeks improved two-point discrimination and touch perception in individuals with ulnar/median nerve damage. More importantly, the authors found that improvements were retained for more than four weeks after the intervention ended. Collectively, this suggests that the release of tonic inhibition on weak muscle pathways, through temporary deafferentation, can lead to functional benefits that are retained long-term.

The Investigators' pilot findings indicate that temporary deafferentation shows similar benefits in the population of SCI. Specifically, it was observed that a single 30-minute session of temporary deafferentation to the stronger biceps can improve excitability to the weaker triceps and result in gains in hand dexterity and pinch strength in SCI.

The Investigators now seek to optimize the current study protocol before a large-scale clinical trial is conducted.

ELIGIBILITY:
Inclusion Criteria:

SCI Patients:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged between 18 and 75 years old
* Have physician diagnosed cervical incomplete spinal cord injury or lesion (iSCI)
* Classified by the American Spinal Cord Association (AIS) impairment scale as AIS C or D
* iSCI occurred at least 18 months ago
* Level of injury or lesion is between C2 and T1
* Bicep strength must be classified as ≥ 3 muscle grade as defined by the medical research council scale
* Tricep strength must be at least an MRC grade of 2 and bet at least 1 muscle grade lower than the bicep
* Both the biceps and triceps will be required to elicit an active motor evoked potential >200 uV with transcranial magnetic stimulation
* Must maintain current medication regime
* Must present with a weaker side of the body, as indicated by a Upper extremity motor score difference between the left and right side
* UEMS < 40 (50 max score)
* Must be able to perform reaching movement training task

Healthy Controls:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged between 18 and 75 years old
* Must be right-handed
* Must be able to perform hand exercises

Exclusion Criteria:

SCI Patients:

* Pacemaker or another implanted device
* Metal in the skull
* History of seizures
* Pregnancy
* First-degree relative with medication-resistant epilepsy
* Current participation in upper limb rehabilitation therapies
* Current use of illicit drugs, abusing alcohol, or have withdrawn from alcohol in the last 6 months
* Other neurological impairment or condition
* Pressure ulcers
* Significant lower motor neuron loss at C7 as noted by a nerve conduction velocity <50 m/s
* History of traumatic brain injury as documented by Rancho Scale Impairment of <5
* History of brain MRI documented focal cerebral cortex infarct (e.g. hydrocephalus)
* Contractures at the elbow
* Severe spasticity as noted by a modified ashworth scale (MAS) > 4
* Documented, non-sedated post-traumatic amnesia lasting more than 48 hours
* Pregnancy
* Allergic to lidocaine
* A neuroactive medication that has the potential to lower the seizure threshold

  * Based on documented publications in stroke, this will include bupropion (wellbutrin), psychostimulants and neuroleptics
  * All medications will be reviewed with physician, Dr. Amol Utturkar (DHR)

Healthy Controls:

* Pacemaker or other implanted device
* Metal in the skull
* History of seizures
* First-degree relative with medication-resistant epilepsy
* Current use of illicit drugs (including heroin, crack/cocaine, marijuana), abusing alcohol or having withdrawn from alcohol in the last 6 months
* Allergy to lidocaine
* Other neurological impairment or condition
* Pregnancy
* A neuroactive medication that has the potential to lower the seizure threshold
* Based on documented publications on stroke, this will include bupropion (wellbutrin), psychostimulants and neuroleptics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2026-06-04 (Estimated); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
Electromyography (EMG) | Throughout Study Duration, an average of four weeks
  The investigators will use an electrical stimulator to send an electrical signal to a target muscle to initiate contraction, and an Electromyography (EMG) will be used to record the changes in target muscle response from baseline, pre-test, and post-test.
  An electronic nerve stimulator will output a pulse ranging from 0 mV to 2 mV for an appropriate maximum muscle contraction to occur, and an Electromyography (EMG in root mean square) will capture the muscle's contraction via surface electrodes. A greater number of Root Mean Square (RMS) millivoltage registered on the EMG signifies a higher response from the muscle, additionally, any plateau of the RMS while administering higher mV from the Stimulator will signify a maximum contraction of the muscle.
Transcranial Magnetic Stimulation (TMS) | Throughout Study Duration, an average of four weeks
  Using Transcranial Magnetic Stimulation (TMS) to promote Motor Evoked Potentials (MEP), the Investigators will monitor changes in cortical excitability of the target muscle's motor hotspot by measuring the muscle excitability with Electromyography (EMG; in millivolts) from Baseline, Pre-test, and at Post-test.
  The motor hotspot of the weak muscle will be defined as the site that evokes MEPs ≥50 mV at the lowest intensity (% device output), or the resting motor threshold (RMT). A decrease of the TMS's percentage output to promote MEPs of the weak muscle signifies a decrease in the cortical excitability, as measured by Active Motor Thresholds (AMT) and Active Motor Evoked Potentials (AMEP).

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Baker, Principal Investigator — University of Texas Rio Grande Valley
Locations (1):
- University of Texas Rio Grande Valley, Harlingen, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data may be shared with interested researchers upon request. There is not a formal sharing plan in place.